CLINICAL TRIAL: NCT00947271
Title: HIV Prevention for STD Clinic Patients
Brief Title: Reducing Sexual Risk Behaviors and Improving Health for People at a Sexually Transmitted Infection Clinic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Rochester (Other); Brown University (Other); Syracuse University (Other)
Responsible Party: Principal Investigator, Michael P. Carey, Director, Centers for Behavioral and Preventive Medicine, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R01MH068171-06 (NIH); R01MH068171-06 (NIH); PCC: DAHBR 9A-ASPQ
Record Dates: First submitted 2009-07-27; First posted 2009-07-28 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: HIV; Sexually Transmitted Diseases; HIV Infections
Keywords: STD; STI; Sexual Behavior; Prevention; HIV seronegativity
MeSH Terms: conditions — Sexually Transmitted Diseases; HIV Infections; Sexual Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- DVD 1 plus assessment 1 (Experimental): Participants will view educational DVD 1 and complete the first version of the study assessment.
  Interventions: Behavioral: DVD 1
- DVD 1 plus assessment 2 (Experimental): Participants will view educational DVD 1 and complete the second version of the study assessment.
  Interventions: Behavioral: DVD 1
- DVD 2 plus assessment 1 (Experimental): Participants will view educational DVD 2 and complete the first version of the study assessment.
  Interventions: Behavioral: DVD 2
- DVD 2 plus assessment 2 (Experimental): Participants will view educational DVD 2 and complete the second version of the study assessment.
  Interventions: Behavioral: DVD 2

INTERVENTIONS:
Behavioral: DVD 1 — The first version of a 20-minute educational DVD aimed to help adult patients reduce sexual risk behaviors (i.e., number of partners, unprotected sex, incident sexually transmitted diseases [STDs]) and improve health
  Arms: DVD 1 plus assessment 1; DVD 1 plus assessment 2
Behavioral: DVD 2 — The second version of a 20-minute educational DVD aimed to help adult patients reduce sexual risk behaviors (i.e., number of partners, unprotected sex, incident STDs) and improve health
  Arms: DVD 2 plus assessment 1; DVD 2 plus assessment 2

SUMMARY:
This study will determine whether showing an educational DVD to people at sexually transmitted infection clinics can reduce incidence of new infections and risky sexual behaviors and improve overall health.

DETAILED DESCRIPTION:
Sexually transmitted infections (STIs) can produce long-term health problems. They are often linked to HIV, which can also be sexually transmitted, because both occur in the same populations and because STIs and HIV interact biologically. Having an STI other than HIV can increase the risk of HIV acquisition and transmission as well as negatively impact HIV progression. The population of people who go to clinics specializing in STIs are particularly at risk of engaging in risky sexual behaviors and having poor health outcomes-like infection with an STI. This study will test the effectiveness of using an educational DVD to reduce incidence of risky sexual behaviors and STI acquisition, including risk of HIV, and to improve overall health.

Participation in this study will involve two phases. In Phase 1, participants will complete both computerized and paper surveys and watch an educational DVD. The educational DVD may include information on diet, physical activity, sleep, smoking, STIs, and stress. Participants will be recruited from among people who are already going to the clinic, and participation will add approximately 1.5 hours to their visits. In Phase 2, participants will be asked to complete four follow-up visits occurring 3, 6, 9, and 12 months after Phase 1. During these follow-up visits, participants will complete a 45-minute computerized survey similar to that in Phase 1 and provide urine and throat samples for STI testing. All surveys will assess health-related thoughts, feelings, and behaviors, including sexual behaviors. Participants will be compensated for completing Phase 1 and each visit in Phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of sexual risk behavior, defined as either signs, symptoms, or diagnosis indicative of an STD during the past 3 months; or unprotected vaginal or anal intercourse with two or more sexual partners, a partner with two or more partners, an anonymous partner, an injection drug using partner, or a partner with an STD

Exclusion Criteria:

* Impaired mental status that would prevent participant from providing informed consent or participating meaningfully
* Inability to understand English

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2009-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Carey, Ph.D., Principal Investigator — The Miriam Hospital and Brown University
Locations (1):
- Monroe County Health Department, Rochester, New York, United States

REFERENCES:
- [Background] Carey MP, Senn TE, Coury-Doniger P, Urban MA, Vanable PA, Carey KB. Optimizing the scientific yield from a randomized controlled trial (RCT): evaluating two behavioral interventions and assessment reactivity with a single trial. Contemp Clin Trials. 2013 Sep;36(1):135-46. doi: 10.1016/j.cct.2013.06.019. Epub 2013 Jun 29. PMID 23816489
- [Derived] Carey KB, Senn TE, Walsh JL, Scott-Sheldon LA, Carey MP. Alcohol Use Predicts Number of Sexual Partners for Female but not Male STI Clinic Patients. AIDS Behav. 2016 Jan;20 Suppl 1(0 1):S52-9. doi: 10.1007/s10461-015-1177-9. PMID 26310596
- [Derived] Carey MP, Senn TE, Walsh JL, Coury-Doniger P, Urban MA, Fortune T, Vanable PA, Carey KB. Evaluating a Brief, Video-Based Sexual Risk Reduction Intervention and Assessment Reactivity with STI Clinic Patients: Results from a Randomized Controlled Trial. AIDS Behav. 2015 Jul;19(7):1228-46. doi: 10.1007/s10461-014-0960-3. PMID 25433653

RESULTS

PARTICIPANT FLOW:
Period: 3 Months Post Intervention
Arm/Group | DVD 1 Plus Assessment 1 | DVD 1 Plus Assessment 2 | DVD 2 Plus Assessment 1 | DVD 2 Plus Assessment 2
Started | 254 | 252 | 254 | 250
Completed | 202 | 204 | 218 | 206
Not Completed | 52 | 48 | 36 | 44
Period: 6 Months Post Intervention
Arm/Group | DVD 1 Plus Assessment 1 | DVD 1 Plus Assessment 2 | DVD 2 Plus Assessment 1 | DVD 2 Plus Assessment 2
Started | 254 | 252 | 254 | 250
Completed | 199 | 199 | 196 | 196
Not Completed | 55 | 53 | 58 | 54
Period: 9 Months Post Intervention
Arm/Group | DVD 1 Plus Assessment 1 | DVD 1 Plus Assessment 2 | DVD 2 Plus Assessment 1 | DVD 2 Plus Assessment 2
Started | 254 | 252 | 254 | 250
Completed | 184 | 192 | 193 | 191
Not Completed | 70 | 60 | 61 | 59
Period: 12 Months Post Intervention
Arm/Group | DVD 1 Plus Assessment 1 | DVD 1 Plus Assessment 2 | DVD 2 Plus Assessment 1 | DVD 2 Plus Assessment 2
Started | 254 | 252 | 254 | 250
Completed | 183 | 192 | 195 | 188
Not Completed | 71 | 60 | 59 | 62

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DVD 1 Plus Assessment 1 | DVD 1 Plus Assessment 2 | DVD 2 Plus Assessment 1 | DVD 2 Plus Assessment 2 | Total
Number analyzed (Participants) | 254 | 252 | 254 | 250 | 1010
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.9 (8.9) | 29.3 (9.7) | 28.0 (9.2) | 28.9 (10.0) | 28.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 100 | 129 | 107 | 443
  Male | 147 | 152 | 125 | 143 | 567
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 2 | 2 | 8
  Asian | 0 | 1 | 3 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2 | 0 | 4
  Black or African American | 168 | 180 | 177 | 166 | 691
  White | 49 | 43 | 43 | 54 | 189
  More than one race | 18 | 14 | 23 | 17 | 72
  Unknown or Not Reported | 16 | 11 | 4 | 11 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 16 | 17 | 24 | 82
  Not Hispanic or Latino | 229 | 236 | 237 | 225 | 927
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 254 | 252 | 254 | 250 | 1010

OUTCOME MEASURES:

1. Primary Outcome: Number of Sexual Partners, 3 Months Post Intervention
Description: number of sexual partners in the past 3 months, assessed 3 months post intervention
Time Frame: Measured after 3 months
Measure: Least Squares Mean (Standard Error); unit: number of partners
Arm/Group | DVD 1 Plus Assessment 1 | DVD 1 Plus Assessment 2 | DVD 2 Plus Assessment 1 | DVD 2 Plus Assessment 2
Number analyzed (Participants) | 202 | 204 | 218 | 206
number of partners | 2.19 (.13) | 2.04 (.11) | 2.14 (.10) | 2.13 (.10)

2. Secondary Outcome: Sexually Transmitted Infection Incidence
Description: number of participants diagnosed with a new STI (CT, Gc, trichomoniasis, syphilis, or HIV) throughout the entire year of follow-up; includes participants who provided a study urine sample for STI testing at 3, 6, 9, and/or 12 months post intervention and participants who received STI testing through the clinic during the year of follow up
Time Frame: Measured throughout the 12 months post intervention
Population: Participants who provided a urine sample for STI testing at any study follow up (3, 6, 9, or 12 months) OR who had STI testing performed at the STI clinic during the 12 months post intervention were included in these analyses
Measure: Number; unit: participants diagnosed with any STI
Arm/Group | DVD 1 Plus Assessment 1 | DVD 1 Plus Assessment 2 | DVD 2 Plus Assessment 1 | DVD 2 Plus Assessment 2
Number analyzed (Participants) | 213 | 219 | 229 | 213
participants diagnosed with any STI | 33 | 36 | 46 | 36

3. Primary Outcome: Number of Sexual Partners, 6 Months Post Intervention
Description: number of sexual partners reported in the past 3 months, assessed 6 months post intervention.
Time Frame: 6 months post intervention
Measure: Least Squares Mean (Standard Error); unit: number of partners
Arm/Group | DVD 1 Plus Assessment 1 | DVD 1 Plus Assessment 2 | DVD 2 Plus Assessment 1 | DVD 2 Plus Assessment 2
Number analyzed (Participants) | 199 | 199 | 196 | 196
number of partners | 1.92 (.13) | 2.18 (.13) | 2.18 (.11) | 2.09 (.13)

4. Primary Outcome: Number of Sexual Partners, 9 Months Post Intervention
Description: number of sexual partners in the past 3 months, assessed 9 months post intervention
Time Frame: 9 months post intervention
Measure: Least Squares Mean (Standard Error); unit: number of partners
Arm/Group | DVD 1 Plus Assessment 1 | DVD 1 Plus Assessment 2 | DVD 2 Plus Assessment 1 | DVD 2 Plus Assessment 2
Number analyzed (Participants) | 184 | 192 | 193 | 191
number of partners | 1.98 (.13) | 1.83 (.10) | 2.11 (.12) | 2.04 (.13)

5. Primary Outcome: Number of Sexual Partners, 12 Months Post Intervention
Description: number of sexual partners in the past 3 months, assessed 12 months post intervention
Time Frame: 12 months post intervention
Measure: Least Squares Mean (Standard Error); unit: number of partners
Arm/Group | DVD 1 Plus Assessment 1 | DVD 1 Plus Assessment 2 | DVD 2 Plus Assessment 1 | DVD 2 Plus Assessment 2
Number analyzed (Participants) | 183 | 192 | 195 | 188
number of partners | 1.84 (.10) | 1.78 (.09) | 1.79 (.09) | 1.90 (.10)

ADVERSE EVENTS:
Arm/Group | DVD 1 Plus Assessment 1 | DVD 1 Plus Assessment 2 | DVD 2 Plus Assessment 1 | DVD 2 Plus Assessment 2
Serious Adverse Events (participants affected / at risk) | 0/254 | 0/252 | 0/254 | 0/250
Other Adverse Events (participants affected / at risk) | 0/254 | 0/252 | 0/254 | 0/250

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No